CLINICAL TRIAL: NCT02837874
Title: Comparisons Between Isoperistaltic and Antiperistaltic Gastrojejunostomy in Laparoscopic Distal Gastrectomy, Randomized Prospective Pilot Study
Brief Title: Comparisons Between Isoperistaltic and Antiperistaltic Gastrojejunostomy in Laparoscopic Distal Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Seung Wan Ryu, Director of Gastrointesinal surgery, professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-02-052
Record Dates: First submitted 2016-07-08; First posted 2016-07-20 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Stomach Neoplasms
Keywords: Gastric cancer; gastrojejunostomy; isoperistaltic; antiperistaltic
MeSH Terms: conditions — Stomach Neoplasms | interventions — Antidiarrheals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isoperistaltic (Active Comparator): Same direction of peristalsis between stomach and jejunum, efferent loop of jejunum is located on the distal part of remnant stomach
  Interventions: Procedure: Isoperistaltic
- Antiperistaltic (Experimental): Reverse direction of peristalsis between stomach and jejunum, efferent loop of jejunum is located on the proximal part of remnant stomach
  Interventions: Procedure: Antiperistaltic

INTERVENTIONS:
Procedure: Isoperistaltic — Same direction of peristalsis between stomach and jejunum, efferent loop of jejunum is located on the distal part of remnant stomach
  Arms: Isoperistaltic
Procedure: Antiperistaltic — Reverse direction of peristalsis between stomach and jejunum, efferent loop of jejunum is located on the proximal part of remnant stomach
  Arms: Antiperistaltic

SUMMARY:
Billroth-II (gastrojejunostomy) is one of major option after gastrectomy for gastric cancer. The investigators hypothesized that isoperistaltic anastomosis lead to higher incidence of dumping syndrome but antiperistaltic (anisoperistaltic) anastomosis have relevance to gastric stasis or obstruction. The investigators will assess complications, dumping syndrome and quality of life between isoperistaltic and antiperistaltic after distal gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
Recently, laparoscopic approach has been a option for gastric cancer, especially early gastric cancer. There are growing interest in quality of life in addition to recurrence or survival. There are few report about peristalsis and no report for quality of life according to a direction of peristalsis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma in stomach
* Scheduled as laparoscopic distal gastrectomy (tumor located lower or middle third)
* Planned with gastrojejunostomy after gastrectomy
* Clinical stage T1N0M0 or T2N0M0
* ECOG 0 or 1 (The Eastern Cooperative Oncology Group)
* ASA score class I-III (The American Society of Anesthesiologists)
* patient has given their written informed consent to participate in the study

Exclusion Criteria:

* Simultaneously combined resection of other organ (including cholecystectomy)
* Active other malignancy
* Requiring total gastrectomy
* Chronic inflammatory bowel disease or other chronic disease related to bowel motility
* Uncontrolled diabetes or patients with diabetic complications
* Vulnerable patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Dumping syndrome | 12 months
  Using Sigstad's score

SECONDARY OUTCOMES:
long-term complication | from 1 month to 12 months
  all kind of complication
Total score of quality of life questionnaire | 12 months
  by EORTC questionnaire
Body weight change | 12 months
  for evaluate nutritional status
Surgical complication | within 1 month
  all kind of complication within 1 month
Gastritis | 12 months
  by endoscopic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Seung Wan Ryu, M.D., Ph.D., Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Banerjee A, Ding Y, Mikami DJ, Needleman BJ. The role of dumping syndrome in weight loss after gastric bypass surgery. Surg Endosc. 2013 May;27(5):1573-8. doi: 10.1007/s00464-012-2629-1. Epub 2012 Dec 12. PMID 23233009
- [Result] Bergamaschi R, Arnaud JP, Marvik R, Myrvold HE. Laparoscopic antiperistaltic versus isoperistaltic gastrojejunostomy for palliation of gastric outlet obstruction in advanced cancer. Surg Laparosc Endosc Percutan Tech. 2002 Dec;12(6):393-7. doi: 10.1097/00129689-200212000-00002. PMID 12496544
- [Result] Mine S, Sano T, Tsutsumi K, Murakami Y, Ehara K, Saka M, Hara K, Fukagawa T, Udagawa H, Katai H. Large-scale investigation into dumping syndrome after gastrectomy for gastric cancer. J Am Coll Surg. 2010 Nov;211(5):628-36. doi: 10.1016/j.jamcollsurg.2010.07.003. Epub 2010 Sep 15. PMID 20829078
- [Result] Houghton AD, Liepins P, Clarke S, Mason R. Iso- or antiperistaltic anastomosis: does it matter? J R Coll Surg Edinb. 1996 Jun;41(3):148-51. PMID 8763175